CLINICAL TRIAL: NCT07006545
Title: Prospective, Multicenter Study of Clinical Rehabilitation and Return-to-activity After Total Knee Arthroplasty
Brief Title: Return to Activity After Total Knee Arthroplasty
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Alexander Franz, Dr. med., B.Sc., University Hospital, Bonn
Other Study IDs: 2024_I
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total Knee Arthroplasty: Patients receiving a total knee arthroplasty
  Interventions: Other: Return to Activity Battery

INTERVENTIONS:
Other: Return to Activity Battery — The main target parameters are muscle mass (sonography), muscle strength (isometric maximum strength measurement), neuromuscular activation (surface EMG), functionality (e.g. 6MWT, chair rising test), knee swelling and subjective assessment of everyday and leisure activities, quality of life (e.g. SF-36) and return to work

SUMMARY:
This multicenter research project aims to correlate objective testing of muscle mass, muscle strength, neuromuscular activation, walking speed and other functional tests with everyday activity and subjective quality of life after total knee arthroplasty. For this purpose, 400 patients from 5 orthopedic departments in Germany and USA will be examined at the time points pre-op, six weeks, three, six and 12 months post-op.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a total knee arthroplasty
* Ability to perform the return to activity battery

Exclusion Criteria:

* Inability to perform the return to activity battery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end-stage gonarthrosis, who have received a total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Muscle Mass | Pre-OP to 12 months Post-OP
  Sonographically Analysis of the M. quadriceps femoris
Muscle Strength | Pre-OP to 12 Months Post-OP
  Isometric maximal strength of the knee extensors

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Technical University Munich, Munich, Bavaria
  - University Hospital Bonn, Bonn, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No